CLINICAL TRIAL: NCT03342053
Title: An Open-Label Extension Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO7234292 (ISIS 443139) in Huntington's Disease Patients Who Participated in Prior Investigational Studies of RO7234292 (ISIS 443139)
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO7234292 (ISIS 443139) in Huntington's Disease Patients Who Participated in Prior Investigational Studies of RO7234292 (ISIS 443139)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BN40697
Record Dates: First submitted 2017-10-31; First posted 2017-11-14 (Actual); Results first posted 2021-01-19 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease | interventions — tominersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- RO7234292 Monthly (Experimental): RO7234292 is administered every 28 days intrathecally for 14 months.
  Interventions: Drug: RO7234292 (RG6042)
- RO7234292 Bimonthly (Experimental): RO7234292 is administered every 56 days intrathecally for 14 months following 2 monthly doses to serve as a loading dose.
  Interventions: Drug: RO7234292 (RG6042)

INTERVENTIONS:
Drug: RO7234292 (RG6042) — Intrathecal injection
  Other Names: Tominersen

SUMMARY:
This study will test the safety, tolerability, pharmacokinetics and pharmacodynamics of RO7234292 administered intrathecally to adult patients with Huntington's Disease.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have completed dosing in ISIS 443139-CS1

Key Exclusion Criteria:

* Any new condition or worsening of existing condition that could make the patient unsuitable for participation or interfere with the patient participating in and/or completing the study

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- The University of British Columbia; The Centre for Huntington Disease, Vancouver, British Columbia, Canada
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Campus Charité Mitte; Klinik für Psychiatrie und Psychotherapi, Berlin
  - St. Josef and St. Elisabeth GmbH ; Klinikum Bochum, Zentralapotheke, Bochum
  - Universitaetsklinikum Ulm, Ulm
- United Kingdom (5):
  - NIHR Welcome Trust Birmingham CRF - University Hospitals Birmingham; Department of Neuropsychiatry, Birmingham
  - University of Cambridge - John van Geest Centre for Brain Repair, Cambridge
  - Cardiff University School of Medicine; Institute of Psychological Medicine Clinical Neurosciences, Cardiff
  - Leonard Wolfson Experimental Neurology Centre, London
  - Central Manchester University Hospitals NHS Foundation Trust; Manchester Centre for Genomic Medicine, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant eligibility for the study was determined within 4 weeks prior to participant entry into the Treatment Period.
Groups:
- RO7234292 Monthly: RO7234292 was administered intrathecally every 28 days for 14 months.
- RO7234292 Bimonthly: RO7234292 was administered intrathecally every 56 days for 14 months following 2 monthly doses to serve as a loading dose.
Period: Overall Study
Arm/Group | RO7234292 Monthly | RO7234292 Bimonthly
Started | 23 | 23
Completed | 21 | 22
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RO7234292 Monthly | RO7234292 Bimonthly | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 20 | 43
  >=65 years | 0 | 3 | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.7 (9.3) | 49.5 (11.3) | 48.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 15 | 13 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 23 | 23 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: One participant's race is known, was reported but cannot be classified in Roche database
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 22 | 23 | 45
    More than one race | 0 | 0 | 0
    Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events
Description: Adverse Events include Adverse Events that started at or after Date/Time of First Exposure to Treatment and procedure-related Adverse Events occurring before the start of treatment.
Time Frame: From baseline up to 18 months
Population: Safety population comprising all participants that were randomized and received at least one dose of RO7234292.
Measure: Number; unit: Percentage of participants
Arm/Group | RO7234292 Monthly | RO7234292 Bimonthly
Number analyzed (Participants) | 23 | 23
Percentage of participants | 100 | 95.7

2. Secondary Outcome: RO7234292 CSF Trough Concentrations by Study Day Prior to Monthly and Bimonthly IT Administration of 120 mg RO7234292 (Primary Analysis)
Time Frame: From baseline to Day 421
Population: CSF Trough Concentrations were reported following study drug administration. Data for Bi-monthly arm was not collected on days 57, 113, 169, 225, 281, 337, 393. Here "Number Analyzed" represents number of participants from whom samples were collected and analyzed.
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | RO7234292 Monthly | RO7234292 Bimonthly
Number analyzed (Participants) | 23 | 23
ng/mL
  Day 29: number analyzed (Participants) | 22 | 21
  Day 29 | 2.59 [1.31 to 12.7] | 2.52 [0.817 to 7.85]
  Day 57: number analyzed (Participants) | 22 | 0
  Day 57 | 3.47 [1.43 to 19.2] |
  Day 85: number analyzed (Participants) | 22 | 21
  Day 85 | 3.70 [1.38 to 7.34] | 1.39 [0.164 to 5.74]
  Day 113: number analyzed (Participants) | 22 | 0
  Day 113 | 3.97 [1.96 to 16.4] |
  Day 141: number analyzed (Participants) | 21 | 21
  Day 141 | 4.57 [1.72 to 13] | 1.35 [0.396 to 3.69]
  Day 169: number analyzed (Participants) | 22 | 0
  Day 169 | 4.47 [2.04 to 12.7] |
  Day 197: number analyzed (Participants) | 21 | 21
  Day 197 | 4.58 [1.74 to 8.61] | 1.26 [0.281 to 3.37]
  Day 225: number analyzed (Participants) | 21 | 0
  Day 225 | 5.21 [1.63 to 14.3] |
  Day 253: number analyzed (Participants) | 20 | 20
  Day 253 | 4.96 [1.56 to 11.8] | 1.45 [0.417 to 3.76]
  Day 281: number analyzed (Participants) | 18 | 0
  Day 281 | 4.96 [1.30 to 12.4] |
  Day 309: number analyzed (Participants) | 18 | 21
  Day 309 | 5.53 [1.74 to 11.6] | 1.35 [0.195 to 2.77]
  Day 337: number analyzed (Participants) | 15 | 0
  Day 337 | 5.12 [2.17 to 10.5] |
  Day 365: number analyzed (Participants) | 18 | 21
  Day 365 | 4.50 [1.18 to 13.9] | 1.45 [0.507 to 2.95]
  Day 393: number analyzed (Participants) | 17 | 0
  Day 393 | 3.10 [0.220 to 9.83] |
  Day 421: number analyzed (Participants) | 18 | 21
  Day 421 | 3.01 [0.239 to 9.54] | 1.34 [0.325 to 2.45]

3. Secondary Outcome: CSF mHTT Protein Concentration Logarithmic Value Change in Geometric Mean (95%CI) From Baseline
Description: The results of the planned analysis related to mHTT protein levels in CSF are reported
Time Frame: From Baseline to Day 421
Population: ITT Population. The data for Bi-monthly arm was not collected on days 113, 169, 225, 281, 337, 393. Here "Number Analyzed" represents number of participants from whom samples were collected and analyzed
Measure: Geometric Mean (95% Confidence Interval); unit: Log (10) fmol/L
Arm/Group | RO7234292 Monthly | RO7234292 Bimonthly
Number analyzed (Participants) | 23 | 23
Log (10) fmol/L
  Day 29: number analyzed (Participants) | 19 | 23
  Day 29 | -27.95 [-38.37 to -15.76] | -21.84 [-33.22 to -8.52]
  Day 57: number analyzed (Participants) | 23 | 2
  Day 57 | -26.90 [-40.95 to -9.50] | 10.11 [-41.68 to 107.88]
  Day 85: number analyzed (Participants) | 22 | 23
  Day 85 | -50.30 [-59.00 to -39.75] | -32.63 [-44.31 to -18.50]
  Day 113: number analyzed (Participants) | 22 | 0
  Day 113 | -49.11 [-58.77 to -37.18] |
  Day 141: number analyzed (Participants) | 22 | 23
  Day 141 | -54.02 [-61.05 to -45.72] | -41.76 [-50.59 to -31.35]
  Day 169: number analyzed (Participants) | 22 | 0
  Day 169 | -42.33 [-53.66 to -28.23] |
  Day 197: number analyzed (Participants) | 22 | 23
  Day 197 | -40.79 [-52.59 to -26.05] | -36.48 [-48.99 to -20.89]
  Day 225: number analyzed (Participants) | 22 | 0
  Day 225 | -47.01 [-58.69 to -32.02] |
  Day 253: number analyzed (Participants) | 21 | 22
  Day 253 | -43.63 [-55.39 to -28.77] | -41.06 [-53.19 to -25.78]
  Day 281: number analyzed (Participants) | 19 | 0
  Day 281 | -40.29 [-58.63 to -13.80] |
  Day 309: number analyzed (Participants) | 18 | 23
  Day 309 | -36.67 [-50.11 to -19.60] | -40.82 [-52.37 to -26.46]
  Day 337: number analyzed (Participants) | 16 | 0
  Day 337 | -42.71 [-58.93 to -20.07] |
  Day 365: number analyzed (Participants) | 19 | 23
  Day 365 | -49.55 [-62.02 to -32.98] | -55.07 [-65.46 to -41.57]
  Day 393: number analyzed (Participants) | 18 | 0
  Day 393 | -41.55 [-59.46 to -15.74] |
  Day 421: number analyzed (Participants) | 19 | 23
  Day 421 | -45.45 [-56.21 to -32.03] | -41.51 [-52.22 to -28.39]

4. Secondary Outcome: Mean Percentage Change in Ventricular Volume Boundary Shift Integral From Baseline to 15 Months
Time Frame: Baseline up to 15 months
Population: Here "Number of Participants Analyzed" represents number of participants from whom data were collected and analyzed. Only data that passed the QC imaging process were included in the analysis.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | RO7234292 Monthly | RO7234292 Bimonthly
Number analyzed (Participants) | 20 | 18
Percentage change | 46.09 (32.14) | 18.77 (10.36)

5. Secondary Outcome: Mean Percentage Change in Caudate Volume Boundary Shift Integral From Baseline to 15 Months
Time Frame: Baseline up to 15 months
Population: Here "Number of Participants Analyzed" represents number of participants from whom data were collected and analyzed.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | RO7234292 Monthly | RO7234292 Bimonthly
Number analyzed (Participants) | 22 | 18
Percentage change | 8.64 (6.26) | 5.67 (2.22)

6. Secondary Outcome: Mean Percentage Change in Whole Brain Volume Boundary Shift Integral From Baseline to 15 Months
Time Frame: Baseline up to 15 months
Population: Here "Number of Participants Analyzed" represents number of participants from whom data were collected and analyzed.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | RO7234292 Monthly | RO7234292 Bimonthly
Number analyzed (Participants) | 13 | 18
Percentage change | 1.63 (1.41) | 0.89 (0.92)

7. Secondary Outcome: EEG Parameters: Mean Change From Baseline to 15 Months in Absolute Power [8-12Hz]
Time Frame: Baseline to 15 Months
Measure: Mean (Standard Deviation); unit: log10(mircrovolts^2)
Arm/Group | RO7234292 Monthly | RO7234292 Bimonthly
Number analyzed (Participants) | 17 | 19
log10(mircrovolts^2) | 0.11 (0.18) | 0.02 (0.21)

8. Secondary Outcome: Mean Change From Baseline in Huntington's Disease Cognitive Assessment Battery Composite Score
Description: HD Cognitive Assessment Battery (HD-CAB) was developed to assess cognitive dysfunction in late premanifest and early manifest HD patients. HD-CAB combines scores from six cognitive tests: SDMT, Self-Paced Tapping, Emotional Recognition, CANTAB One Touch Stocking, Hopkins Verbal Learning Test - Revised, and Trail-Making Test. A multi-component score is derived by transforming the subject's score on each cognitive test to a z-score. Using z-scores permits the combination of test scores with different scales. Unlike other measures that use an external reference population to create z-scores, HD-CAB uses the baseline data of the study. Individually, for each of the six cognitive tests, the study baseline mean is subtracted from the subject's score, and this value is divided by the study baseline standard deviation. The six z-scores are averaged to produce the HD-CAB score. A positive change from baseline indicates improvement in cognitive function; a negative change indicates worsening.
Time Frame: Baseline to 15 Months
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | RO7234292 Monthly | RO7234292 Bimonthly
Number analyzed (Participants) | 17 | 21
z-score | -0.33 (0.27) | -0.15 (0.23)

ADVERSE EVENTS:
Time Frame: From baseline to up to 18 months
Description: Safety population comprising all participants that were randomized and received at least one dose of RO7234292
Arm/Group | RO7234292 Monthly | RO7234292 Bimonthly
All-Cause Mortality (participants affected / at risk) | 1/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 4/23 | 3/23
Other Adverse Events (participants affected / at risk) | 22/23 | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RO7234292 Monthly (N=23) | RO7234292 Bimonthly (N=23)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Myelitis (Infections and infestations) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meningitis chemical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Hyporeflexia (Nervous system disorders) | 1 (1) | 0 (0)
Neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RO7234292 Monthly (N=23) | RO7234292 Bimonthly (N=23)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 5 (6)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (5)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 3 (3) | 1 (1)
Gait disturbance (General disorders) | 6 (14) | 0 (0)
Injection site pain (General disorders) | 2 (3) | 4 (4)
Puncture site pain (General disorders) | 2 (3) | 2 (4)
Ear infection (Infections and infestations) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 9 (14) | 10 (15)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 1 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (4)
Contusion (Injury, poisoning and procedural complications) | 6 (21) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 18 (87) | 12 (17)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 4 (10) | 5 (6)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 2 (4)
Procedural pain (Injury, poisoning and procedural complications) | 7 (19) | 12 (15)
Skin abrasion (Injury, poisoning and procedural complications) | 7 (11) | 4 (6)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
CSF protein increased (Investigations) | 2 (3) | 1 (1)
CSF white blood cell count increased (Investigations) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (6) | 2 (2)
Balance disorder (Nervous system disorders) | 3 (3) | 1 (1)
Cerebral ventricle dilatation (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Dysarthria (Nervous system disorders) | 2 (3) | 0 (0)
Dyskinesia (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 6 (13) | 4 (10)
Hyperkinesia (Nervous system disorders) | 2 (2) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 2 (2) | 0 (0)
Motor dysfunction (Nervous system disorders) | 3 (3) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Parkinsonism (Nervous system disorders) | 2 (2) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Depressed mood (Psychiatric disorders) | 2 (2) | 2 (2)
Depression (Psychiatric disorders) | 4 (4) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2)
Irritability (Psychiatric disorders) | 2 (3) | 0 (0)
Tension (Psychiatric disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Haematoma (Vascular disorders) | 4 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT03342053/Prot_SAP_000.pdf